CLINICAL TRIAL: NCT07141992
Title: Comparison of Active vs Passive Neural Mobilizations Effects in Improving Burning Pain, Muscular Strength, and Range of Motion in Patients With Diabetic Neuropathy: A Randomized Control Trial
Brief Title: Comparison of Active vs Passive Neural Mobilizations Effects in Improving Burning Pain, Muscular Strength, and Range of Motion in Patients With Diabetic Neuropathy
Acronym: RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: Baqai Institute of Diabetology and Endocrinology (Other)
Responsible Party: Principal Investigator, MUHAMMAD MEHRAN HAIDER, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB No. 3966
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Neuropathy; Diabete Mellitus; Diabetic Neuropathy
Keywords: Active Neural mobilizations; Passive Neural mobilizations; diabetic neuropathy; neuropathic pain; muscle strength improvement; ROM improvement; pain reduction
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of Active Neural Mobilization on Pain, Strength, and ROM in Diabetic Neuropathy (Experimental): Participants in the active neural mobilization group will receive neural flossing techniques, aimed at improving nerve mobility and reducing neuropathic symptoms. Along with neural mobilization, participants will follow a standardized physiotherapy protocol, including:
  Gait training on both smooth and rough surfaces Strengthening exercises: leg press, ankle press, isometric exercises for knee and ankle extensors, bridging, and pelvic rolling All exercises will be performed in 3 sets of 12 repetitions, with 30 seconds of rest between sets Stationary cycling will be included as part of cardiovascular conditioning The intervention will be delivered over 12 sessions, scheduled three times per week for four weeks. This program aims to reduce burning pain, and enhance muscle strength and range of motion in patients with diabetic neuropathy.
  Interventions: Other: Active Neural Mobilzations
- Effect of Passive Neural Mobilization on Pain, Strength, and ROM in Diabetic Neuropathy (Experimental): Participants in the passive neural mobilization group will receive neural tensioning techniques, which involve therapist-guided passive movements to mobilize the neural structures. In addition to passive mobilization, participants will undergo the same standardized physiotherapy protocol, which includes:
  Gait training on both smooth and rough surfaces Strengthening exercises: leg press, ankle press, isometric exercises for knee and ankle extensors, bridging, and pelvic rolling Exercises will be performed in 3 sets of 12 repetitions, with 30 seconds of rest between sets Stationary cycling will be used for cardiovascular conditioning This group will also receive 12 treatment sessions, conducted three times per week over four weeks, with the goal of improving pain, strength, and mobility in individuals with diabetic neuropathy.
  Interventions: Other: Passive Neural Mobilzations

INTERVENTIONS:
Other: Active Neural Mobilzations — Participants in this group will receive active neural mobilization in the form of neural flossing techniques. These involve controlled, repeated movements performed actively by the patient to mobilize peripheral nerves without placing them under excessive tension. The goal is to restore neural mobility, reduce mechanosensitivity, and relieve neuropathic symptoms such as burning pain.
  Arms: Effect of Active Neural Mobilization on Pain, Strength, and ROM in Diabetic Neuropathy
Other: Passive Neural Mobilzations — Participants in this group will receive passive neural mobilization using neural tensioning techniques. These techniques involve therapist-applied passive limb movements that place a controlled tensile load on the neural structures. The objective is to improve neural gliding, reduce nerve compression, and decrease neuropathic pain, particularly in cases of restricted neural tissue mobility.
  Arms: Effect of Passive Neural Mobilization on Pain, Strength, and ROM in Diabetic Neuropathy

SUMMARY:
* Randomized controlled trial evaluating active and passive neurodynamic techniques for diabetic neuropathy.
* Sample size: 60 patients (30 per group), aged 40 to 65 years, diagnosed with diabetes mellitus.
* Exclusion criteria: Systemic diseases, pregnancy, fractures, foot ulceration, amputation, osteoarthritis.
* Study will be conducted at physiotherapy OPDs of Dow Ojha Hospital, DIPMR,NIDE and Baqai Institute of Diabetology and Endocrinology.
* Participants randomly assigned into two groups using a computer-generated randomization sheet.

Group A: Active neurodynamics (neural flossing) - patient-controlled nerve gliding movements.

Group B: Passive neurodynamics (tensioners) - therapist-applied nerve stretches.

* Standard treatment includes gait training, lower limb strengthening exercised, and stationary bike sessions.
* Treatment: 12 sessions over 4 weeks (3 sessions per week, 30 minutes each session).
* Assessments will be done at baseline and post-intervention by a blinded physical therapist.
* Outcome measures: DN-4 (pain), MMT (muscle strength), Goniometry (ROM), LLTT (nerve mobility).
* Data were analyzed using SPSS Version 27. A one-way ANOVA was performed to compare the results before and after the intervention.
* Study duration: 9 months, including approval, pilot study, data collection, and final presentation.
* Study aims to determine the most effective neurodynamic technique for pain relief, mobility, and muscle strength.
* Findings will guide better rehabilitation strategies for improved patient outcomes and quality of life.

DETAILED DESCRIPTION:
Diabetic neuropathy is a common complication of diabetes mellitus that presents with neuropathic pain, muscle weakness, and restricted mobility in the lower limbs. These impairments negatively affect quality of life and increase the risk of falls, foot ulcers, and amputations. Pharmacological treatments are available but frequently provide incomplete symptom relief and may cause adverse effects, creating the need for effective non-pharmacological interventions.

Neural mobilization techniques have been reported to improve nerve mobility and decrease pain sensitivity. Two forms will be applied in this trial: active neural mobilization (neural flossing) and passive neural mobilization (tensioners). Both approaches aim to restore normal neural dynamics but differ in their application principles.

This randomized controlled trial will be conducted in the physiotherapy outpatient departments of Dow Ojha Hospital, the National Institute of Diabetology and Endocrinology (NIDE), and the Baqai Institute of Diabetology and Endocrinology (BIDE). A total of 60 participants with clinically diagnosed diabetic neuropathy, aged 40-65 years, will be recruited and randomly assigned to either an active neural mobilization group or a passive neural mobilization group.

Each group will receive 12 treatment sessions over a 4-week period. Both groups will additionally perform conventional physiotherapy, including gait training, strengthening exercises, and stationary cycling. Outcomes will be assessed at baseline and post-intervention. Measures will include:

Neuropathic pain using the DN-4 questionnaire

Muscle strength using manual muscle testing (MMT)

Joint range of motion using goniometry

The primary objective of the study will be to compare the effectiveness of active versus passive neural mobilization in reducing neuropathic pain and improving muscle strength and joint mobility. Secondary objectives will include determining clinical applicability and the potential role of these interventions in rehabilitation protocols for diabetic neuropathy.

Limitations of the trial will include the inability to blind participants, possible variability in treatment adherence, and potential influence of external factors such as concurrent analgesic use. Randomization and standardized intervention protocols will be employed to minimize bias.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female individuals
* Aged between 40 and 65 years
* Diagnosed with Diabetes Mellitus (Type I and Type II)
* Diagnosis confirmed by a physician

Exclusion Criteria:

* One with any systemic disease
* Medical conditions (neurological disorders, fractures, acute inflammatory conditions, recent surgeries)
* Foot Ulceration
* Amputation
* OA of Ankle or Knee Joint

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Lower Limb Tension Test | 12 sessions for 4 weeks
  Lower Limb Tension Test (LLTT) Purpose: Assess neural mechanosensitivity of lower limb nerves, especially sciatic, tibial, and peroneal nerves.
  Also Known As: Straight Leg Raise (SLR), Slump Test, Prone Knee Bend Test, etc.
  Indications:
  Radiating leg pain Suspected lumbar radiculopathy Neural tension syndromes
  Procedure Includes:
  Hip flexion, knee extension, ankle dorsiflexion, and/or foot inversion/eversion based on nerve bias
  Positive Sign:
  Reproduction of neuropathic symptoms (burning, tingling, shooting pain) Symptoms change with sensitizing maneuvers
  Used In:
  Neuropathy Sciatica Disc herniation Piriformis syndrome
DN-4 (Douleur Neuropathique en 4 questions) | 12 sessions in 4 weeks
  DN-4 Questionnaire (Douleur Neuropathique en 4 questions) Purpose: To screen for neuropathic pain and distinguish it from nociceptive pain.
  Total Items: 10 7 sensory descriptors (e.g., burning, electric shocks, tingling, numbness) 3 clinical examination findings (e.g., hypoesthesia to touch or pinprick, pain on brushing)
  Scoring:
  Each "yes" = 1 point Total Score Range: 0 to 10 Score ≥ 4 indicates likely neuropathic pain Time Required: Less than 5 minutes
  Advantages:
  Quick and easy to administer Non-invasive High sensitivity and specificity
  Used In:
  Diabetic neuropathy Post-stroke pain
  Sciatica
  Postherpetic neuralgia
Goniometery (Joint Range of Motion) | 12 sessions for 4 weeks
  Goniometry Purpose: Measure joint range of motion (ROM) accurately Instrument: Goniometer (standard)
  Components:
  Axis: Placed over the joint Stationary arm: Aligned with proximal segment Moving arm: Aligned with distal segment
  Procedure:
  Explain to patient → Proper positioning → Stabilize proximal joint → Move limb through ROM → Read measurement
  Used To Assess:
  Joint mobility limitations Effectiveness of treatment Progress tracking in rehabilitation Common Areas: Knee, hip, ankle, shoulder, elbow, wrist, cervical spine
Manual Muscle Testing | 12 sessions in 4 weeks
  Manual Muscle Testing (MMT) Purpose: Evaluate muscle strength manually
  Grading Scale (0-5):
  0 = No contraction
  1. = Flicker/trace of contraction
  2. = Full ROM in gravity-eliminated position
  3. = Full ROM against gravity
  4. = Full ROM with some resistance
  5. = Full ROM with maximum resistance (normal)
  Procedure:
  Proper positioning → Isolate target muscle → Apply resistance gradually → Grade based on performance
  Used In:
  Neuromuscular conditions Orthopedic rehab Stroke, SCI, peripheral nerve injuries
  Advantages:
  Quick and cost-effective Useful in baseline assessment and progress monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Ishaque Khan, PhD, Study Director — Dow Institute of Physical Medicine and Rehabilitation, Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences / Baqai Institute of Diabetology and Endocrinology, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to confidentiality concerns. Protecting the privacy and anonymity of participants is a top priority, and sharing IPD may risk breaching this confidentiality. Additionally, the data is securely stored and intended solely for use within the scope of this study; therefore, it will not be shared with other researchers.

REFERENCES:
- [Background] Goyat M, Saxena A, Goyal M. Study Protocol titled as "Effectiveness of neural mobilization in improving the ankle ROM and plantar pressure distribution in patients with diabetic peripheral neuropathy: A single group, pre post, quasi experimental study protocol". J Diabetes Metab Disord. 2022 Aug 15;21(2):2035-2041. doi: 10.1007/s40200-022-01106-z. eCollection 2022 Dec. PMID 36404825
- See also: Study Protocol titled as "Effectiveness of neural mobilization in improving the ankle ROM and plantar pressure distribution in patients with diabetic peripheral neuropathy: A single group, pre post, quasi experimental study protocol" — https://pubmed.ncbi.nlm.nih.gov/36404825/
- See also: Effects of foot and ankle mobilisations combined with home stretches in people with diabetic peripheral neuropathy: a proof-of-concept RCT — https://pubmed.ncbi.nlm.nih.gov/38057930/
- See also: Effects of Neural Mobilization in Diabetic Peripheral Neuropathy: A Scoping Review — https://pubmed.ncbi.nlm.nih.gov/38205228/